CLINICAL TRIAL: NCT06000306
Title: Measurable Residual Disease Monitoring by Digital Droplet PCR in the Early Period After Allogeneic Hematopoietic Stem Cell Transplantation to Predict Patients at High Risk of Relapse
Brief Title: MRD Monitoring by Digital Droplet PCR in the Early Period After Allo-HSCT to Predict Patients at High Risk of Relapse
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, He Huang, The President of The First Affiliated Hospital, College of Medicine, Zhejiang University, Zhejiang University
Other Study IDs: IIT20230588C-R1
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Measurable Residual Disease
Keywords: droplet digital PCR; allogeneic hematopoietic stem cell transplantation; relapse
MeSH Terms: conditions — Neoplasm, Residual; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ddPCR MRD positivity
  Interventions: Diagnostic Test: Digital Droplet PCR
- ddPCR MRD negativity
  Interventions: Diagnostic Test: Digital Droplet PCR

INTERVENTIONS:
Diagnostic Test: Digital Droplet PCR — Measurable residual disease Monitoring by Digital Droplet PCR in the Early Posttransplant Period

SUMMARY:
A study on the Effectiveness of digital droplet PCR in monitoring measurable residual disease during the early period after allogeneic hematopoietic stem cell transplantation to predict patients at high risk of relapse

DETAILED DESCRIPTION:
This is a retrospective and multicenter clinical study.This study is indicated for patients with hematological malignancies who underwent allo-HSCT. It aims to evaluate the effectiveness of digital droplet PCR in monitoring measurable residual disease during the early period after allogeneic hematopoietic stem cell transplantation to predict patients at high risk of relapse. 192 patients will be enrolled. The clinical end points include cumulative incidence of relapse, relapse-free survival, non-relapse mortality, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. The presence of at least one haematological tumour-associated mutation or fusion gene detected at diagnosis by NGS or real-time qPCR provided for posttransplant MRD monitoring;
2. Successful stem cell engraftment
3. Received at least one bone marrow MRD detection by ddPCR in +30 days to +120 days after HSCT;
4. Age 12-70

Exclusion Criteria:

1. Patients who relapsed or died before the first ddPCR monitoring;
2. Patients with only germline mutations.

Ages: 12 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hematological malignancies who underwent allo-HSCT were enrolled for MRD mornitoring in the early period of allo-HSCT
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of relapse (CIR) | At Year 2
  The time from the date of transplantation to disease recurrence:
  Disease recurrence, defined as one of the following:
  Leukemia blasts reappeared in peripheral blood, or blasts ≥ 5%, naive monocytes ≥ 5% in bone marrow, or extramedullary lesions.

SECONDARY OUTCOMES:
Relapse-free survival (RFS) | At Year 2
  The time from the date of treatment to the occurrence of any of the following:
  1. Death from any cause
  2. Disease recurrence
Non-relapse mortality (NRM) | At Year 2
  Assessment of NRM at Year 2
Overall survival (OS) | At Year 2
  Assessment of OS at Year 2

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Zhejiang Medical Colleage Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Chen W, Huang J, Zhao Y, Huang L, Yuan Z, Gu M, Xu X, Shi J, Luo Y, Yu J, Lai X, Liu L, Fu H, Bao C, Huang X, Zheng Z, Huang H, Hu X, Zhao Y. Measurable residual disease monitoring by ddPCR in the early posttransplant period complements the traditional MFC method to predict relapse after HSCT in AML/MDS: a multicenter retrospective study. J Transl Med. 2024 Apr 30;22(1):410. doi: 10.1186/s12967-024-05114-w. PMID 38689269